CLINICAL TRIAL: NCT00034281
Title: A Phase I, Open-Label, Dose Escalating, Multiple Dose Study to Determine the Safety, Tolerability, Maximum Tolerated Dose and Pharmacokinetics of Oral TAK-165 Administered Once Daily to Subjects With Tumors Known to Express HER2.
Brief Title: Safety and Tolerability Study of TAK-165 in Subjects With Tumors Expressing HER2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-01-TL-165-001; U1111-1127-6123 (Registry Identifier: WHO)
Record Dates: First submitted 2002-04-24; First posted 2002-04-25 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Breast Neoplasm; Pancreatic Neoplasm; Lung Neoplasm; Ovarian Neoplasm; Renal Neoplasm
Keywords: Gene, HER2; Clinical Trial, Phase I; Breast neoplasm; Pancreatic neoplasm; Ovarian neoplasm; Colorectal neoplasm; Renal neoplasm; Prostate neoplasm; Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Kidney Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Neoplasms | interventions — TAK-165

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-165 QD (Experimental)
  Interventions: Drug: TAK-165

INTERVENTIONS:
Drug: TAK-165 — Starting dose of TAK-165 10 mg, tablets, orally, once daily with dose escalation to tolerability for 56 days.

SUMMARY:
The purpose of this study is to investigate a safe dose of TAK-165, once daily (QD), in patients with HER2-tumor expression.

DETAILED DESCRIPTION:
The human epidermal growth factor receptor 2 (HER2) is a member of the Type 1 family of growth factor tyrosine kinases. HER2 forms hetero- and homo-dimers with other members of this family of tyrosine kinases. As a result of dimerization at the cell surface, intracellular signal transduction is initiated, resulting in cell proliferation.

HER2 expression has been observed in a variety of human tumors including breast cancer, non-small cell lung cancer, prostate cancer, pancreatic cancer, renal cell cancer, and ovarian cancer. HER2 overexpression is associated with clinically more aggressive breast cancer, and is an independent predictor of poor prognosis in patients with breast cancer.

TAK-165 is an active and selective inhibitor of tyrosine kinase activity of HER2 being developed for patients with lower levels of HER2 expression. This study will seek to determine the safety, tolerability, maximum tolerated dose and pharmacokinetics of TAK-165 administered to subjects with tumors known to express HER2.

The total duration of the study will be at minimum 8 weeks, or 56 Days. Subjects without progressive disease after 8 weeks may continue to receive study drug, provided that they do not meet criteria for withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Have advanced or metastatic cancer which is refractory to standard therapy or subjects for whom there is no known effective therapy.
* Have a histologically or cytologically proven diagnosis of a solid tumor known to express HER2.
* Have a predicted life expectancy of greater than or equal to 12 weeks.
* Have a Karnofsky Performance Status of greater than or equal to 60%
* Have recovered from toxicities of prior chemotherapy, surgery, or radiotherapy.

Exclusion Criteria:

* Be pregnant or lactating. Women of childbearing potential must have a negative serum pregnancy test result within 7 days of enrollment into the study. Male and female subjects of childbearing potential (including women who have been amenorrheic for less than 1 year) must use appropriate birth control during the entire duration of the study, or the subject must be surgically sterile.
* Have symptomatic brain metastasis
* Have received any other anti-cancer treatment or investigational drug/treatment within 28 days prior to study Day 1.
* Have a history of another malignancy within the last 5 years.
* Have inadequate organ function.
* Have heart failure defined by an ejection fraction of less than or equal to 50% as measured by MUGA.
* Have Class II, III or IV symptoms of heart failure as defined by the New York Heart Association, or uncontrolled arrhythmias, or recent history of myocardial infarction or angina pectoris.
* Have a medical condition that may interfere with intake and/or absorption of the study drug (e.g., gastrectomy or resection of major portion of small intestine).
* Have any other serious disease or condition present at screening or at study Day 1 that might affect life expectancy or make it difficult to successfully manage and follow the subject according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-06; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Days 8, 15, 22, 28 and every 14 days thereafter to Final Visit
Maximum Tolerated Dose | Days 8, 15, 22, 28 and every 14 days thereafter to Final Visit
Optimal Dosing for Phase II Studies. | End of Study.

SECONDARY OUTCOMES:
Clinical Pharmacokinetic Profile of TAK-165 | Days 8, 15, 22, 28 and every 14 days thereafter to Final Visit
Response Evaluation Criteria in Solid Tumors Documentation of Objective Tumor Response. | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (4):
- United States (4):
  - Arizona Cancer Center, Scottsdale, Arizona
  - The Institute for Drug Development, San Antonio, Texas
  - Brooke Army Medical Center/Drug Development Unit, San Antonio, Texas
  - South Texas VA, Audie Murphy Division, San Antonio, Texas